CLINICAL TRIAL: NCT03405207
Title: Vitamin D Deficiency Treatment Outcomes on Inflammation, Endothelial Function and Ventricular Retrieval After Non ST-Segment Elevation Myocardial Infarction: A Randomized Placebo Controlled Clinical Trial (NAVID Study)
Brief Title: Vitamin D Deficiency Treatment Outcomes After Non-ST-Segment Elevation Myocardial Infarction
Acronym: NAVID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Masoumeh Sadeghi, Dr. Masoumeh Sadeghi, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Isfahan Vitamin D Non-ST-MI
Record Dates: First submitted 2018-01-07; First posted 2018-01-23 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Vitamin D Deficiency; Non-ST Elevation Myocardial Infarction (nSTEMI); Inflammation; Coronary Artery Disease With Myocardial Infarction
MeSH Terms: conditions — Vitamin D Deficiency; Non-ST Elevated Myocardial Infarction; Inflammation; Coronary Artery Disease, Autosomal Dominant, 1 | interventions — Bulk Drugs

STUDY DESIGN:
Intervention Model Description: we have 2 groups entitled active drug receiver and placebo receiver and patients will randomly allocated between these two groups at first and continue until finishing the study.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active drug receiving group (Active Comparator): the drug is vitamin D3 50000 UNT oral capsule prescribing under Holick's protocol, which is every week for 8 weeks then every month for long life
  Interventions: Drug: Vitamin D3 50000 UNT Oral Capsule
- placebo receiving group (Placebo Comparator): the same as active comparator unless the drug is the identical placebo oral capsule
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Vitamin D3 50000 UNT Oral Capsule — Holick's protocol of treating vitamin D deficiency lasting for 8 weeks
  Other Names: active drug
  Arms: active drug receiving group
Drug: Placebo oral capsule — identical as active drug providing by pharmaceutical company unless it is placebo
  Other Names: placebo
  Arms: placebo receiving group

SUMMARY:
The leading cause of death in the world is due to cardiovascular events, which originate from coronary artery stenosis therefore it affects myocardial blood flow and finally may cause infarction. Atherosclerosis is the most debatable hypothesis in coronary stenosis. Scientists think body inflammation is one of the main etiologies. There are many factors affect this inflammatory process, which Vitamin D is one of them. Vitamin D deficiency has been linked to various inflammatory diseases. However, the mechanism by which vitamin D reduces inflammation remains poorly understood. Vitamin D deficiency is pandemic around the world with 30-50% prevalence in adult population and several evidences advocated its association with immune-based disease. Additionally, there are some study suggesting patients who suffered from myocardial infarction have lower serum vitamin D level. It has been revealed Vitamin D deficiency has numerous major drawbacks on cardiovascular system. Its deficiency benefits atherosclerosis progression and may cause endothelial inflammation and dysfunction in coronary artery. There is not any evidences study vitamin D deficiency treatment on non ST-Segment Elevation Myocardial Infarction nor there is any study demonstrating its effect on cardiovascular health through Holick's protocol. Furthermore endothelial function, cardiac work retrieval and inflammation after 8 weeks has not been studied with this protocol yet.

According to current data, the investigators assume by treating this vital and worldwide deficit in our body, doctors can help decrease inflammation, decelerate the atherosclerosis progression and enhance ventricular function after infarction.

Besides all of the recognized risk factors, vitamin D deficiency should be considered a very important and mischievous cardiovascular alarm for the body, which should be treated and maintained through the whole life due to lack of sufficient sunlight exposure and nutrition intake.

In preventive medicine domain, the investigators anticipate by maintaining a high level of this vitamin in the body, cardiovascular events decrease and its burden on society will decline to much extend leading to a higher quality of life and health worldwide.

DETAILED DESCRIPTION:
The leading cause of death in the world is due to cardiovascular events, which originate from coronary artery stenosis therefore it affects myocardial blood flow and finally may cause infarction. ST-Segment elevation is an indicator of infarction (STEMI) in electrocardiography (ECG) besides cardiac enzymes like troponin; however, there is another type of infarction without elevation, which called non ST-Segment Elevation myocardial infarction (NSTEMI).

The most established method of treating this condition is percutaneous coronary intervention (PCI) and balloon angiography although in some cases coronary artery bypass grafting surgery is more beneficial. Atherosclerosis is the most debatable hypothesis in coronary stenosis. Scientists think body inflammation is one of the main etiologies. There are many factors affect this inflammatory process, which Vitamin D is one of them. Vitamin D deficiency has been linked to various inflammatory diseases. However, the mechanism by which vitamin D reduces inflammation remains poorly understood. Vitamin D Inhibits Monocyte/Macrophages Pro-inflammatory Cytokine Production by Targeting mitogen-activated protein kinase (MAPK) Phosphatase-1 and nuclear factor kappa-light-chain-enhancer of activated B cells (NF-κB) pathway therefore decrease production of IL-6 and tumor necrosis factor-alpha (TNFα) and increasing interleukin (IL) 10 and transforming growth factor beta (TGFβ) from human monocytes. Chronic inflammatory diseases that are vitamin D deficient (20 ng/ml) may benefit from oral supplementation of vitamin D to get their serum vitamin D level>30 ng/ml.

Galectin-3 is emerging fibrotic biomarkers that is thought to be causally involved in the development of heart failure. Galectin-3 is a beta-galactoside binding lectin that is produced by macrophages during myocardial stress and activates fibroblasts. Besides its roles in inflammation and in cellular adhesion, galectin-3 plays an important role in cardiac fibrosis. Furthermore, galectin-3 has an established role as a modulator in tumor progression. Galectin-3 is released in the circulation, and can be measured reliably and has been shown to independently predict outcomes in heart failure patients and in the general population. However, galectin-3 is not cardiac specific, but is expressed in several fibrotic and inflammatory diseases.

Vitamin D is one of the fat-soluble micronutrients, which sunlight is the principle key to make this vitamin in our body. Vitamin D deficiency is pandemic around the world with 30-50% prevalence in adult population and several evidences advocated its association with immune-based disease like asthma, multiple sclerosis (MS), Type 2 diabetes and many cancers. Additionally, there are some study suggesting patients who suffered from myocardial infarction have lower serum vitamin D level. It has been revealed Vitamin D deficiency has numerous major drawbacks on cardiovascular system. Its deficiency benefits atherosclerosis progression and may cause endothelial inflammation and dysfunction in coronary artery. Endothelial malfunction with lipid sedimentation beneath the intima layer attract leukocytes and make foam cells. Therefore it leads to produce active agents and make smooth muscle cells to proliferate and lead the lumen to be narrower, which consequently decrease oxygenated blood flow and causes ischemia and infarction. Monocyte chemoattractant protein 1 (MCP-1) and n-terminal fragment of pro-brain natriuretic peptide (NT-pro-BNP) are two newly discovered molecules associated independently with coronary calcification level. MCP-1 has a role in representing the relationship between acute myocardial infarction and inflammation.

Renin-Angiotensin-Aldosterone system has a principle role in blood pressure maintenance. It has been shown this vitamin can regulate this system too.

Hypocalcemia in vitamin D deficiency activate parathyroid gland to produce parathormone (PTH), which makes bones to release calcium and kidneys to reabsorb calcium from urine more. PTH activates the α1-hydroxylase of the Kidney to produce activated vitamin D (calcitriol or 1,25(OH)2 VitD) from stored-form (cholecalciferol or 25(OH) VitD). Calcium is the leading cation in the cardiac myocyte which contributes in contraction, contractility and voltage conduction. Also phosphorous excrete more due to PTH effect on distal convoluted tubule. Alkaline phosphatase is an indicator of bone metabolism in resorbing the hydroxyapatite crystals. Body regulate the level of phosphorous by fibroblasts growth factor (FGF) 23 and PTH accurately. FGF-23 is secreted by osteocytes in response to elevated calcitriol. FGF-23 decreases the reabsorption and increases excretion of phosphate in Kidneys. FGF-23 may also suppress α1-hydroxylase, reducing its ability to activate vitamin D and subsequently impairing calcium absorption. It has been shown in some studies that FGF-23 level was independently associated with endothelial function, arterial stiffness, vascular calcification, ventricular hypertrophy, renal failure progression, and cardiovascular related mortality. Similarly, PTH level has the same relationship. In conclusion, these studies proposed vitamin D deficiency has a major role in endothelial dysfunction, inflammation, myocardial infarction and stroke.

FGF21 has lately emerged as a potent metabolic regulator with multiple effects that ultimately improve the lipoprotein profile. Early studies show that FGF21 is associated with the presence of atherosclerosis and may play a protective role against plaque formation by improving endothelial function.

High level of Homocysteine which is one of the amino acids metabolism end products, make the patient to be more susceptible to endothelial cell injury which therefore make inflammation and atherosclerosis and finally ischemia. Hyperhomocysteinemia is therefore a risk factor for coronary artery disease. In one randomized controlled trial (RCT) involving 3096 patients who referred for PCI treated with a combination of Vitamin B 6, 9 and 12 and suggested although these vitamins has a lot of major effects in biochemical metabolism and antioxidant action, hospital readmission and re-infarction was not decreased. This study was just the beginning of the new era in managing cardiovascular events by controlling its biological risk factors.

PRIMO trial of 196 participants who had renal failure and left ventricular hypertrophy consumed an analog of activated vitamin D called paricalcitol and assessed left atrial volume index after 24 and 48 weeks. This trial had come to an end and had a lot of problems including they study population, type of drug they chose, co-founder variables and lack of sufficient follow up. To follow this field, VITDAMI trial ameliorate the PRIMO problems and investigate the effects of consuming 0.266 milligrams calcifediol each 2 weeks in 144 acute anterior STEMI patients on left ventricular remodeling using cardiac magnetic resonance imaging (MRI) and assessing its left ventricular end diastolic volume (LV-EDV) after 1 year. Its result has not been published yet. To power up their study, they will evaluate endothelial function, calcium metabolism products and aspects of inflammation. Calcifediol is produced by the liver enzyme 25-hydroxylase from its pro-hormone cholecalciferol (Vitamin D3), and its blood concentration is considered the best indicator of vitamin D status. Although there are several vitamin D deficiency treatment protocol, using calcifediol is not prevalent worldwide. Holick et al. demonstrated a type of protocol in which the patient with hypovitaminosis D (25(OH) Vitamin D less than 20 ng/ml) received 50,000 international units (IU) of Vitamin D3 or D2 (Cholecalciferol or Ergocalciferol respectively) once a week for 8 weeks to achieve calcifediol levels higher than 30 ng/ml then continue on maintenance dose (50,000 IU every month or 1,500-2,000 IU/day) for the rest of the life. This procedure has been tolerated well by patients and has high acceptance rate. One study compared Holick's method with another common protocol and established there were no difference in increasing the serum level of vitamin D nor patients' preference.

In the CANTHOS study, the anti-IL-1β antibody prescribed in three different doses for patients with established atherosclerosis and high level of C-reactive protein (CRP) and follow them up to 48 months and evaluated nonfatal myocardial infarction, nonfatal stroke, or cardiovascular death. They suggested the anti-inflammatory effects of canakinumab led to a significantly lower rate of recurrent cardiovascular events at a dose of 150 mg every 3 months. For the first time, in this RCT, which the most valuable methodology in medical investigations and causality evaluations, the investigators will evaluate one of the most prevalent management protocols of vitamin D deficiency (Holick's) on one of the most dramatic human disease which obtained the higher burden of disease worldwide, myocardial infarction. There is currently only one evidence studying the effects of consuming calcifediol on anterior ST-Segment Elevation Myocardial Infraction. the investigators decided to choose a different drug (cholecalciferol) with different approach and different MI (NSTEMI). In this study the investigators will use no invasive instruments and assessing controversial variables outcomes to open a big door to cardiovascular disease management and preventive medicine to much extend.

ELIGIBILITY:
Inclusion Criteria:

1. 30-65 years old patients
2. Hypovitaminosis D (serum 25(OH) Vitamin D< 20 ng/ml)
3. Written and informed consent to participate in this project
4. Non ST-Segment Elevation Myocardial Infarction: any patients with chest pain or any discomfort and suspected MI who referred to our Heart Center Emergency Room without any ST-Segment Elevation (according to J-point) in 12-lead ECG (according to American Heart Association (AHA) guidelines) plus increasing level of serum cardiac Troponin I

Exclusion Criteria:

1. Normal Vitamin D level
2. Body mass index (BMI)>30 kg/m2
3. Do not tend to attend in this study
4. Any life-threatening medical condition
5. Hyperparathyroidism (parathyroid hormone (PTH)>upper normal limit according to lab reference range)
6. Liver failure (any positive past medical history or Aspartate and Alanine aminotransferase (AST and ALT) 2 times more than normal upper limit)
7. Renal Failure (any positive past medical history or Glomerular filtration rate <60 ml/min/1.73 m2 estimated with MDRD formula of Qx calculate application)
8. Any prior history of diagnosed cancer, rheumatologic and immunologic disorders

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
endothelial function(1) change from baseline | change from baseline at 8th weeks after infarction
  E-Selectin of blood
endothelial function(2) change from baseline | change from baseline at 8th weeks after infarction
  fibroblast growth factor 21 of blood
endothelial function(3) change from baseline | change from baseline at 8th weeks after infarction
  fibroblast growth factor 23 of blood
endothelial function(4) change from baseline | change from baseline at 8th weeks after infarction
  vascular cell adhesion molecule 1 of blood
endothelial function(5) change from baseline | change from baseline at 8th weeks after infarction
  inter-cellular cell adhesion molecule 1 of blood
endothelial function(6) change from baseline | change from baseline at 8th weeks after infarction
  with flow mediated dilation (FMD)

SECONDARY OUTCOMES:
inflammation state(1) changes from baseline | change from baseline at 8th weeks after infarction
  C-reactive protein (CRP) of blood
ventricular function(1) changes from baseline | change from baseline at 8th weeks after infarction
  galectin-3 of blood
inflammation state(2) changes from baseline | change from baseline at 8th weeks after infarction
  monocytes chemo attractant protein-1 (MCP-1) of blood
inflammation state(3) changes from baseline | change from baseline at 8th weeks after infarction
  interleukin 10 of blood
inflammation state(4) changes from baseline | change from baseline at 8th weeks after infarction
  interleukin 6 of blood
inflammation state(5) changes from baseline | change from baseline at 8th weeks after infarction
  transforming growth factor beta (TGF-β) of blood
ventricular function(2) changes from baseline | change from baseline at 8th weeks after infarction
  n-terminal of brain natriuretic peptide of blood
ventricular function(3) changes from baseline | change from baseline at 8th weeks after infarction
  echocardiography assessing ejection fraction (EF%)
ventricular function(4) changes from baseline | change from baseline at 8th weeks after infarction
  echocardiography assessing left ventricular end diastolic volume
ventricular function(5) changes from baseline | change from baseline at 8th weeks after infarction
  doing strain echocardiography for changes of heart function in stress situations

CONTACTS AND LOCATIONS:
Overall Officials: masoumeh sadeghi, M.D., Principal Investigator — Cardiac Rehabilitation Research Center, Isfahan Cardiovascular Research Institute
Locations (1):
- Cardiovascular Rehabilitation Research Center, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No